CLINICAL TRIAL: NCT00338559
Title: Does Using Laryngeal Mask Airway (LMA) Instead of an Endotracheal Tube (ET Tube) Affect the Incidence of Postoperative Vomiting in Children Undergoing Strabismus Correction? - An Observational Study
Brief Title: Does LMA Instead of ET Tube Affect Incidence of Postoperative Vomiting in Children Undergoing Strabismus Correction?
Status: Completed | Type: Observational
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Samia Khalil, Professor - Anesthesiology, The University of Texas Health Science Center, Houston
Other Study IDs: HSC-MS-06-0059
Record Dates: First submitted 2006-06-15; First posted 2006-06-20 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Strabismus
Keywords: Strabismus; LMA; ET Tube; POV
MeSH Terms: conditions — Strabismus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- LMA group: Patients in which laryngeal mask airway (LMA) is used.
- ET group: Patients in which endotracheal tube (ET) is used.

SUMMARY:
The effect of airway management on vomiting after strabismus surgery is unknown. The purpose of this study is to find out whether the use of different airway devices, such as LMA, which is a special mask placed in the throat or Endotracheal tube (ET tube), which is a soft tube placed in the wind pipe, affects the incidence of vomiting after surgery. Two hundred six children between the ages of 2 and 12 years are expected to take part in this study.

DETAILED DESCRIPTION:
The child will be checked by the study doctor to determine if he/she qualifies to be part of the study. The study doctor may not want the child to take part in this study if he/she is currently in another research study; or if the child has been in any other research study within the last 30 days, or if the child is extremely obese, or has reflux or another GI problem.

If the child qualifies for the study, he/she will receive routine general anesthesia. For airway management, the child will have either a LMA or ET tube. The child has an equal chance of receiving either one of these airways devices, much like the coin flip.

After surgery, the child will be transferred to the recovery room (PACU). If the child vomits in PACU, he/she will receive rescue medication, which can be repeated if the need arises.

A research coordinator will call the parents the following day to find out whether the child vomited after leaving the hospital, in the car or at home, for any complications and receiving any medications.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Elective Uni- or Bilateral Strabismus repair

Exclusion Criteria:

* ASA >2
* History of Prematurity
* History of Reflux
* History of Neurological Disease
* Difficult Airway
* Obesity

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Two hundred six children between the ages of 1 and 12 years are expected to take part in this study.
Sampling Method: Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2006-05; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Numbers of the patients that will develop postoperative vomiting in children undergoing strabismus correction | 2 days

CONTACTS AND LOCATIONS:
Overall Officials: Samia N Khalil, MD, Principal Investigator — University of Texas HSC at Houston
Locations (1):
- Memorial Hermann Hospital, Houston, Texas, United States